CLINICAL TRIAL: NCT06381271
Title: Transcatheter Aortic Valve Replacement for Pure Severe Aortic Valve Regurgitation: a Real-world, Prospective, Multicenter Study (TRUST TAVR Registry)
Brief Title: Transcatheter Aortic Valve Replacement for Pure Severe Aortic Valve Regurgitation
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: TRUST TAVR Registry
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Regurgitation
Keywords: Aortic Valve Regurgitation; TAVR; Real-Word
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — A total of 500 consecutive patients with NAVR undergoing TAVR will be enrolled at 3-5 centers. Clinical follow-up will be conducted in the periprocedural and after aortic valve implantation at 1 month, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years
  Other Names: Transcatheter aortic valve implantation

SUMMARY:
The purpose of this multicenter, prospective and observational registry is to evaluate the safety and efficacy of TAVR for treatment of pure severe aortic valve regurgitation. Baseline characteristics, procedural and clinical data will be collected

DETAILED DESCRIPTION:
Pure native aortic valve regurgitation (NAVR) is a multifactorial valvular disease, with a prevalence of moderate or severe NAVR ranging from 0.5% to 2.7%. Patients with severe NAVR have a poor prognosis, conservative management has a 1-year mortality rate of more than 20%. Currently, surgical aortic valve replacement (SAVR) is the recommended treatment strategy for patients with NAVR. However, data showed that only 20% of patients with severe NAVR and left-ventricular ejection fraction (LVEF) of 30-50% undergo SAVR, while only 3% of those with an LVEF below 30% receive SAVR. Therefore, a less invasive surgical alternative therapy is needed for high surgical-risk patients from SAVR.

Transcatheter aortic valve replacement (TAVR) is now considered the first-choice treatment for elderly patients with aortic stenosis, regardless of surgical risk. Recently, it has also been used to treat patients with NAVR in an "off-label" setting. The latest European guidelines suggest that TAVR may be considered in experienced centers for selected patients with AR who are not eligible for SAVR. However, the role of TAVR in patients with severe NAVR is still debatable. Current studies on this topic are limited by their retrospective design and small sample sizes.

Dedicated devices for aortic regurgitation, such as the JenaValve, have shown promising results in terms of technical success and short-term outcomes. However, TAVR for patients with NAVR using on-label devices has a relatively high rate of pacemaker implantation. Additionally, the dedicated device was designed only for tricuspid valve anatomy, making TAVR with off-label devices the main invasive strategy for high-surgical risk patients with bicuspid valves. It's worth noting that the dedicated device is not yet commercially available worldwide. Therefore, further investigation into TAVR using off-label devices for NAVR patients, including those with bicuspid and tricuspid valves, is necessary.

The objective of this study was to evaluate the safety and efficacy of TAVR in patients with NAVR in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with severe aortic valve regurgitation undergo evaluation by the Heart team and are eligible for TAVR therapy.
* 2. Patients who understand the purpose of this study, agree to participate in the trial and sign the informed consent form

Exclusion Criteria:

* 1. Patients who cannot provide informed consent
* 2. Patients who are treated with TAVR for aortic stenosis
* 3. Patients who are participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pure severe native aortic valve regurgitation underwent TAVR
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2034-10 (Estimated)

PRIMARY OUTCOMES:
Combined clinical efficacy outcomes | 1 year
  Combined clinical efficacy outcomes as composed by all-cause mortality, all strokes, any hospitalization

SECONDARY OUTCOMES:
Combined early safety and clinical efficacy outcomes | 30 days
  Composed by all-cause mortality, all strokes, life-threatening or fatal bleeding, major vascular, access-related, or cardiac structural complication, acute kidney injury stage 3 or 4, moderate or severe aortic regurgitation, new permanent pacemaker due to procedure-related conduction abnormalities, conduction block and arrhythmia, surgery or intervention related to the device, any hospitalization, myocardial infarction, any other adverse events
Rate of technical success | at exit from procedure room
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Rate of device success | discharge or 30 days
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient<20mmHg, and less than moderate aortic regurgitation)
Combined clinical efficacy outcomes | 2 years, 3 years, 4 years
  Combined clinical efficacy outcomes as composed by all-cause mortality, all strokes, any hospitalization
Rate of all-cause mortality | 5years and 10years
Valve-related long-term clinical efficacy | 5 years and 10 years
  * Freedom from bioprosthetic Valve Failure (defined as: Valve-related mortality OR Aortic valve re-operation/re-intervention OR Stage 3 hemodynamic valve deterioration)
  * Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies)
  * Freedom from VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns (e.g. clinically apparent leaflet thrombosis)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D, Ph.D, Study Chair — Xijing Hospital; Rutao Wang, M.D, Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No